CLINICAL TRIAL: NCT06993454
Title: Acute Exercise and Endogenous Glucose Production in Type 2 Diabetes: Implications for Glycemic Control and Treatment of Hepatic Steatosis
Acronym: ACELERATE-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2238850
Record Dates: First submitted 2025-04-11; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Hepatic Steatosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatty Liver

STUDY DESIGN:
Intervention Model Description: This research design is a cross-sectional, parallel trial with two groups: lean, healthy controls and individuals with T2D and hepatic steatosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean, healthy controls (Other): Control group.
  Interventions: Other: Magnetic Resonance Liver Assessment; Other: Bike Exercise VO2max; Other: DEXA
- Individuals with T2D and hepatic steatosis (Other): T2D group.
  Interventions: Other: Magnetic Resonance Liver Assessment; Other: Bike Exercise VO2max; Other: DEXA

INTERVENTIONS:
Other: Magnetic Resonance Liver Assessment — Liver fat will be measured by MR imaging to assess level of hepatic steatosis.
Other: Bike Exercise VO2max — Maximal fitness measured by cycle ergometer.
Other: DEXA — Measure body composition (fat and lean body mass).

SUMMARY:
The overall aim of this study is to investigate the effects of exercise on the amount of glucose that is made by the liver in people with and without Type 2 diabetes (T2D) and hepatic steatosis (fatty liver).

ELIGIBILITY:
Inclusion criteria for individuals with T2D and elevated liver fat ≥5.6%

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or (pre-menopausal) female, aged 25-55 years
4. Body mass index (BMI) between 25 and 45 kg/m2
5. Sedentary (1 day or less per week of structured exercise)
6. Type 2 diabetes mellitus: HbA1c ≥7.5%
7. Liver fat ≥5.6% based on MRI
8. Weight stable (± 2 kg) for prior 3 months

Inclusion criteria for lean, healthy controls

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or (pre-menopausal) female, aged 25-55 years
4. Body mass index (BMI) between 18.5 and 27.5 kg/m2
5. Normal liver fat (FibroScan CAP <249dB/m, <5.6% liver fat based on MRI)
6. Weight stable (± 2 kg) for prior 3 months
7. Active (≥3 day/week of structured exercise)

Exclusion Criteria

1. Exclusion criteria for individuals with T2D and elevated liver fat ≥5.6% Currently taking insulin, incretin mimetics, and/or thiazolidinediones
2. Any change in glucose-lowering medications within the previous three months.
3. Inability to stop any medications which interfere with glucose metabolism for visits 4 and 7.
4. Resting blood pressure ≥ 160/100 mm Hg
5. Triglycerides ≥ 500 mg/dL
6. Any renal, cardiac, liver, lung, or neurological disease that in the opinion of the principal investigator would compromise participant safety or the participants' ability to complete the exercise protocol
7. Any significant disease or unstable medical condition (i.e., coronary heart disease, chronic renal failure, chronic hepatic disease, severe pulmonary disease)
8. Presence of clinically significant abnormalities on electrocardiogram (ECG) that is a contra-indication to exercise testing
9. Cancer (active malignancy with or without concurrent chemotherapy; except for basal cell carcinoma)
10. Pregnancy during the previous 6 months, lactating, or planned pregnancy in the next 6 months
11. Post- or peri-menopausal women
12. Partial and/or full hysterectomy (self-report)
13. Use of drugs known to affect energy metabolism or body weight: including, but not limited to orlistat, sibutramine, ephedrine, phenylpropanolamine, corticosterone, etc
14. Hyperthyroidism including those with normal TSH (0.35-4.5) on pharmacological treatment; individuals with hypothyroidism may be referred to their primary care provider for evaluation and retested; any medication change for hypothyroidism must be stable for ≥3 months prior to retesting
15. Current treatment with blood thinners or anti-platelet medications that cannot be safely stopped for testing procedures
16. New onset (<3 months on a stable regime) hormone replacement therapy
17. Current use of beta-adrenergic blocking agents
18. Major surgery on the abdomen, pelvis, or lower extremities within previous 3 months
19. Previous bariatric or other surgery for obesity
20. Abnormal blood count/anemia (hemoglobin <12 g/dl in men or 11 g/dl in women; Hct <34%), blood transfusion or blood donation within the last 2 months
21. Current smokers (smoking within the past 3 months prior to screening visit, including any/all tobacco products)
22. Current drug or alcohol abuse/dependence, or positive urine toxicology screen
23. Alcohol consumption >7 drinks per week for women or 14 drinks per week for men or history of binge drinking (≥5 drinks for males or 4 drinks for females in a 2-hour period more than once per month)
24. Metal implants (pacemaker, aneurysm clips) based on investigator's judgment at screening
25. Not physically capable of performing the exercise required of the study protocols
26. Unable to participate in Magnetic Resonance Imaging (MRI) assessments due to physical limitations of equipment tolerances (e.g. MRI bore size) based on investigator's judgment at screening.
27. Unable to tolerate MRI or claustrophobia.
28. Diagnosed psychotic or psychiatric conditions prohibiting adherence to study protocol; hospitalization for any psychotic or psychiatric condition within one year
29. Self-reported chronic, active, or latent infection requiring chronic antibiotic or anti-viral treatment; Human Immunodeficiency Virus (HIV); active hepatitis B or C undergoing antiviral therapy
30. Unable or unwilling to communicate with staff or to provide written informed consent

Exclusion criteria for lean, healthy controls

1. Currently taking insulin, injectable incretin mimetics, and/or thiazolidinediones
2. Taking glucose-lowering medications
3. HbA1c ≥ 5.7%; pre-diabetes, type 2 diabetes, or type 1 diabetes
4. Resting blood pressure ≥ 160/100 mm Hg
5. Triglycerides ≥ 500 mg/dL
6. Any renal, cardiac, liver, lung, or neurological disease that in the opinion of the principal investigator would compromise participant safety or the participants' ability to complete the exercise protocol
7. Any significant disease or unstable medical condition (i.e., coronary heart disease, chronic renal failure, chronic hepatic disease, severe pulmonary disease)
8. Presence of clinically significant abnormalities on electrocardiogram (ECG) that is a contra-indication to exercise testing
9. Cancer (active malignancy with or without concurrent chemotherapy; except for basal cell carcinoma)
10. Pregnancy during the previous 6 months, lactating, or planned pregnancy in the next year
11. Post- or peri-menopausal women
12. Partial and/or full hysterectomy (self-report)
13. Use of drugs known to affect energy metabolism or body weight: including, but not limited to orlistat, sibutramine, ephedrine, phenylpropanolamine, corticosterone, etc
14. Hyperthyroidism including those with normal TSH (0.35-4.5) on pharmacological treatment; individuals with hypothyroidism may be referred to their primary care provider for evaluation and retested; any medication change for hypothyroidism must be stable for ≥3 months prior to retesting
15. Current treatment with blood thinners or anti-platelet medications that cannot be safely stopped for testing procedures
16. New onset (<3 months on a stable regime) hormone replacement therapy
17. Current use of beta-adrenergic blocking agents
18. Major surgery on the abdomen, pelvis, or lower extremities within previous 3 months
19. Previous bariatric or other surgery for obesity
20. Increased liver function tests (AST/ALT/GGT/or alkaline phosphatase greater than 2.5 times the upper limit of normal)
21. Abnormal blood count/anemia (hemoglobin <12 g/dl in men or 11 g/dl in women; Hct <34%), blood transfusion or blood donation within the last 2 months
22. Current smokers (smoking within the past 3 months prior to screening visit, including any/all tobacco products)
23. Current drug or alcohol abuse/dependence, or positive urine toxicology screen
24. Alcohol consumption >7 drinks per week for women or 14 drinks per week for men or history of binge drinking (≥5 drinks for males or 4 drinks for females in a 2-hour period more than once per month)
25. Metal implants (pacemaker, aneurysm clips) based on investigator's judgment at screening
26. Not physically capable of performing the exercise required of the study protocols
27. Unable to participate in Magnetic Resonance Imaging (MRI) assessments due to physical limitations of equipment tolerances (e.g. MRI bore size) based on investigator's judgment at screening.
28. Unable to tolerate MRI or claustrophobia.
29. Diagnosed psychotic or psychiatric conditions prohibiting adherence to study protocol; hospitalization for any psychotic or psychiatric condition within one year
30. Self-reported chronic, active, or latent infection requiring chronic antibiotic or anti-viral treatment; Human Immunodeficiency Virus (HIV); active hepatitis B or C undergoing antiviral therapy
31. Unable or unwilling to communicate with staff or to provide written informed consent

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Measurement of Endogenous Glucose Production (EGP) | Day 14
  Bulk EGP will be measured during resting and exercise conditions to determine how Endogenous Glucose Production (EGP) differs during exercise (compared to no exercise) in T2D and Metabolic dysfunction associated steatotic liver disease (MASLD).

CONTACTS AND LOCATIONS:
Overall Officials: Justine Mucinski, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States